CLINICAL TRIAL: NCT01881607
Title: Respiratory Symptoms, Asthma and Passive Smoking in Children: Effectiveness of an Integrated Individual, Family, and School-based Intervention
Brief Title: An Integrated Intervention to Reduce Secondhandsmoke in Children
Acronym: RESPIR·NET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Public Health Agency of Barcelona (Other); Institut Municipal d'Investigació Mèdica (Unknown); Fundació La Marató de TV3 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 040830; 64/04 (Other: Bellvitge's CEIC)
Record Dates: First submitted 2013-06-05; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Secondhand Exposure; Smoking Status
Keywords: tobacco smoke pollution; Tobacco use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Schoolchildren aged 12-13 years in the first year of Compulsory Secondary Education (Enseñanza Secundaria Obligatoria in the Spanish educational system) in the city of Terrassa. The CONTROL arm is formed by schoolchildren in schools that willnot receive the intervention and will continue with ongoing (usual) health education sessions.
- Intervention (Experimental): The intervention at the classroom consisted of six sessions with the pupils of one hour each that were conducted by the teacher/tutor. We provided the teachers with a training session and a teachers' guide, and we gave each pupil a workbook with the activities. At the school level, the intervention consisted of four types of posters with specific messages directed to students, teachers, and parents, and the fourth poster type advertised the new smoking laws. we gave teachers and school managers the guide "Towards a Smoke-Free School" to facilitate the prevention and control of smoking (active and passive) in the school environment. Family level activities: Parents were required to complete the "My risk thermometer" activity at home with their children. Parents received a brochure with information on the risks of SHS exposure and recommendations to prevent SHS exposure, and a refrigerator magnet with the logo of the program.
  Interventions: Behavioral: RESPIRNET Program

INTERVENTIONS:
Behavioral: RESPIRNET Program — The intervention at the classroom consisted of six sessions with the pupils of one hour each that were conducted by the teacher/tutor. We provided the teachers with a training session and a teachers' guide, and we gave each pupil a workbook with the activities. At the school level, the intervention consisted of four types of posters with specific messages directed to students, teachers, and parents, and the fourth poster type advertised the new smoking laws. we gave teachers and school managers the guide "Towards a Smoke-Free School" to facilitate the prevention and control of smoking (active and passive) in the school environment. Family level activities: Parents were required to complete the "My risk thermometer" activity at home with their children. Parents received a brochure with information on the risks of SHS exposure and recommendations to prevent SHS exposure, and a refrigerator magnet with the logo of the program.
  Arms: Intervention

SUMMARY:
This is a community essay to assess the effectiveness of a multi-level (individual, family, and school) school-based intervention to prevent the exposure to secondhand smoke (SHS) in a population of 1,734 schoolchildren (12-14 years old) in Terrassa (Catalonia, Spain). Schools were assigned to the intervention or the controlgroup at random. The investigators assessed SHS exposure in different settings (at school, at home, on transportation and leisure time) and tobacco consumption by means of a questionnaire before and one year after the intervention. Based on a previously evaluated intervention to prevent smoking initiation (PASE/ESFA program) the investigators designed a new intervention (the RESPIR•NET Program) including two new activities to prevent passive smoking to be applied at three levels: in the classroom (pupils), at the school (pupils, teachers, and parents), and in the family (pupils and parents).

ELIGIBILITY:
Inclusion Criteria:

* all schoolchildren attending the school at the day of interview

Exclusion Criteria:

* absence of school
* language problems with questionnaire

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1779 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of exposure to secondhand smoke | 1 year
  The prevalence of exposure to secondhand smoke is computed by dividing the number of children exposed / total number of children. Exposure to secondhand smoke is obtained using a questionnaire at baseline and one year later. The questionnaire was prepared from previously validated questionnaires on SHS.

SECONDARY OUTCOMES:
Prevalence of current smokers | 1 year
  The prevalence of smoking is computed by dividing the number of smoking children / total number of children. Smoker status is obtained using a questionnaire at baseline and one year later. The questionnaire has been previously validated in other investigations.

CONTACTS AND LOCATIONS:
Locations (1):
- Catalan Institute of Oncology, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Martin-Pujol A, Fernandez E, Schiaffino A, Moncada A, Ariza C, Blanch C, Martinez-Sanchez JM; RESPIR.NET research group. Tobacco smoking, exposure to second-hand smoke, and asthma and wheezing in schoolchildren: a cross-sectional study. Acta Paediatr. 2013 Jul;102(7):e305-9. doi: 10.1111/apa.12232. Epub 2013 Apr 16. PMID 23581609
- [Derived] Blanch C, Fernandez E, Martinez-Sanchez JM, Ariza C, Lopez MJ, Moncada A, Schiaffino A, Rajmil L, Salto E, Pascual JA, Nebot M; RESPIR.NET research group. Impact of a multi-level intervention to prevent secondhand smoke exposure in schoolchildren: a randomized cluster community trial. Prev Med. 2013 Nov;57(5):585-90. doi: 10.1016/j.ypmed.2013.07.018. Epub 2013 Aug 7. PMID 23933268